CLINICAL TRIAL: NCT00623844
Title: Prevention Through Acitivity in Kindergarten Trial
Brief Title: Prevention Through Activity in Kindergarten Trial
Acronym: PAKT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Wuerzburg (Other)
Collaborators: Gmünder ErsatzKasse GEK (Unknown); University of Cologne (Other)
Responsible Party: Principal Investigator, Helge Hebestreit, Prof. Dr. med., University of Wuerzburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BMBF 01EL0606
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2014-12

CONDITIONS: Child, Preschool
Keywords: Prevention; Physical activity; Obesity; Motor skills; Kindergarten
MeSH Terms: conditions — Motor Activity; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Physical activity intervention: structured daily 30-min activity classes at preschool, activity homeworks, parent and teacher education
  Interventions: Behavioral: physical activity
- Control (No Intervention): Keep usual activities in kindergarten

INTERVENTIONS:
Behavioral: physical activity — activity program at kindergarten 5 * 30 min per week plus education of parents (letters, flyers, presentations, counselling) plus activity homework for children involving also the families
  Arms: Intervention

SUMMARY:
Objectives: The PAKT project shall evaluate the effects of an exercise intervention in kindergarten combined with an educational training of parents and kindergarten teachers on behavior and health status of children.

Study design: Baseline measurements were performed on more than 700 kindergarten children aged 43-67 months in May to July 2007. The kindergartens are located in and around Wuerzburg in Germany. Kindergartens were then randomized in an intervention (21 kindergartens) and a control (20 kindergartens) group. The intervention group offers a daily exercise class lasting at least 30 min. Parents and teachers of the children in the intervention program receive educational training. In addition, the children have activity homework involving the entire family. The control kindergartens keep their routine. Follow-up measurements of physical activity (actigraph), motor skills, body mass index, skinfold thickness, and blood pressure take place in January/February 2008, June/July 2008, and September/October 2008. The number of accidents in and outside of the kindergartens and the number of children missing the kindergarten due to infections are monitored continuously.

Use of results: If the PAKT program should proof effective, the results will be published in scientific journals and made public using the press. With the help of the GEK, the program will then be implemented nationwide in kindergartens.

ELIGIBILITY:
Inclusion Criteria:

* Children in participating kindergartens

Exclusion Criteria:

* Health conditions restricting physical activity
* Age < 43 months or > 67 months

Ages: 43 Months to 67 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 718 (Actual)
Dates: Start 2007-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Physical activity | baseline, after 4-5 and 8-9 months of intervention, 2-4 months after intervention
  Accelerometry over 7 days
motor skills | baseline, after 4-5 and 8-9 months of intervention, 2-4 months after intervention
  Composite score of several motor tasks

SECONDARY OUTCOMES:
adiposity | baseline, after 4-5 and 8-9 months of intervention, 2-4 months after intervention
  BMI, skinfolds
blood pressure | baseline, after 4-5 and 8-9 months of intervention, 2-4 months after intervention
accidents | baseline, after 4-5 and 8-9 months of intervention, 2-4 months after intervention
infections | baseline, after 4-5 and 8-9 months of intervention, 2-4 months after intervention
television viewing time | baseline, after 4-5 and 8-9 months of intervention, 2-4 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Helge Hebestreit, MD, PhD, Principal Investigator — University of Wuerzburg

REFERENCES:
- [Derived] Roth K, Mauer S, Obinger M, Ruf KC, Graf C, Kriemler S, Lenz D, Lehmacher W, Hebestreit H. Prevention through Activity in Kindergarten Trial (PAKT): a cluster randomised controlled trial to assess the effects of an activity intervention in preschool children. BMC Public Health. 2010 Jul 12;10:410. doi: 10.1186/1471-2458-10-410. PMID 20624316